CLINICAL TRIAL: NCT05508724
Title: An Observational Study of the Relationship Between Pressure-volume Curves and Recruitability of the Lung in Mechanically Ventilated Critically Ill Patients With Respiratory Failure
Brief Title: Recruitment Manoeuvres in Critically Ill Patients
Acronym: RMCIP
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, Dr Jessica Souza Luiz, Research Fellow in Clinical Pulmonary Physiology, University of Oxford
Other Study IDs: PID16097; IRAS 306692 (Other: Health Research Authority NHS UK)
Record Dates: First submitted 2022-07-22; First posted 2022-08-19 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Distress Syndrome; Respiratory Insufficiency; Respiratory Failure; Shock Lung
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically-ill mechanically ventilated patients: Intensive Care patients receiving mechanical ventilation due to respiratory failure

SUMMARY:
Diseases of the lungs can be life-threatening. When these organs fail to adequately work, treatments to support their function are offered, often in Intensive Care Units (ICU). Respiratory failure patients may need sedation and placement of a tube in their windpipe so that a mechanical ventilator can take over their breathing until they have recovered enough to breathe again on their own. One problem that occurs in patients under mechanical ventilation is that parts of the lung tissue tend to collapse (atelectasis), reducing the amount of the lung that is able to transfer oxygen and carbon dioxide effectively and even progressing to pneumonia.

To address this problem, ICU doctors often perform a procedure named 'recruitment manoeuvre', which involves briefly inflating the patient's lungs with enough pressure to try to open up the collapsed areas of lung. However, fundamental aspects of the change in the functioning of the heart and lungs that occur during and after such manoeuvre are not fully understood.

In this study, funded by the University of Oxford, the investigators wish to study patients with respiratory failure who are receiving mechanical ventilation. Participants will be recruited at the ICU of the Royal Berkshire Hospital having their cardiopulmonary data collected over the course of a day. During this period, some patients will be assessed to determine whether they may benefit from a recruitment manoeuvre using a pressure-volume curve. As this assessment is not perfect, the investigators wish to study which features of this curve predict a successful recruitment. The investigators will do this by evaluating the volume of the lung before and after the recruitment manoeuvre is performed using a device named Optical Gas Analyser.

A better understanding of the effects of the recruitment manoeuvre will help the investigators to determine how and when such manoeuvres should be performed in critically ill patients.

DETAILED DESCRIPTION:
Critical care units provide supportive therapies to help patients survive a period of life-threatening illness. Among such treatments, mechanical ventilation constitutes an essential asset to assist in patient recovery from respiratory failure and to provide airway protection in neurologically compromised patients. The need for mechanical ventilation is more often driven by respiratory failure than a need for neuroprotection. In excess of 100,000 adult patients are mechanically ventilated in UK ICUs annually, and this number has risen considerably recently due to the emergence of the COVID-19 pandemic.

Respiratory failure may be triggered by pulmonary (e.g., pneumonia, acute respiratory distress syndrome, interstitial fibrosis) or extra-pulmonary (e.g., sepsis, shock) disturbances. The abnormal function of the cardiorespiratory system in these critical conditions results in carrying degrees of hypoxaemia and hypercapnia, leading to the need for respiratory support by mechanical ventilation.

In patients undergoing mechanical ventilation for respiratory failure, the lung is characterized by a much-enhanced tendency to collapse. This collapse worsens hypoxaemia, and increases the stress and strain applied to those regions of the lung that remain aerated, leading to ventilator-induced lung injury (VILI). Re-aeration of non-aerated lung (recruitment) improves oxygenation and prevents VILI. For this reason, some clinicians employ recruitment manoeuvres following intubation, or subsequently during their ICU stay. However, it remains unclear which patients benefit from this intervention, at what time point(s) it is most beneficial, and the underlying mechanisms.

It is recognised that the volume of lung that is potentially recruitable (recruitability) varies widely from patient to patient, being influenced by: (i) the underlying disease precipitating respiratory failure (pulmonary versus extrapulmonary injury); (ii) the distribution of lung injury (lobar versus non lobar); and (iii) the time from initiation of lung injury.

An ability to assess recruitability is a pre-requisite for a rational recruitment strategy and selecting parameters for mechanical ventilation. The gold standard to assess recruitability involves performing a CT scan at two different levels of inspiratory pressure and assessing the mass of lung tissue (grams) that transitions from a non-aerated to an aerated state. This is not feasible in everyday clinical practice since it is time consuming, requires transfer of a critically ill patient to the radiology suite, and involves a significant exposure to ionising radiation. An alternative is to use some measure of the change in lung volume between the different pressure levels, but this is not the same as a change in non-aerated lung mass and indeed the two measures may not even be correlated.

It has been suggested that certain parameters derived from a low-flow inflation and deflation pressure-volume (PV) curve might be useful in the prediction of lung recruitability. When a sustained inflation recruitment manoeuvre is performed, the increase in volume evident on the curve should theoretically give a measure of the volume recruited during the manoeuvre. Based on a similar PV curve principle, recruitment-to-inflation ratio (RI) was developed as a single-breath assessment of lung recruitability. However, these strategies for the bedside assessment of recruitability have received limited validation and currently provide only a qualitative analysis, whereby the patient's lungs will be considered to have either a high or a low potential of recruitment.

Finally, electric impedance tomography has been advocated by some as an alternative tool to assess recruitment but has not been widely adopted into clinical use.

The decision as to whether or not to perform a recruitment manoeuvre in a given patient currently relies on individual consultant preference and clinical judgement, leading to variation within medical practice. Due to an inadequate understanding of the full physiological effects associated with this intervention, it can be difficult to decide whether lung recruitment is likely to prove useful for a given patient. For example, a recruitment manoeuvre that increases lung volume is more likely to be beneficial if it results in an even inflation of a larger alveolar volume than if it arises purely as an increase in dead space.

To date, there is no consensus regarding recruitment manoeuvres and the existing guidance is limited.

The broad objective of this prospective, observational study is to gain a better understanding of how to predict the effects of recruitment manoeuvres in patients who are being mechanically ventilated for respiratory failure. The opportunity to examine this area more closely than has previously been possible, arises from the development of technology to make highly precise measurements of respiratory exchange non-invasively in these patients: the Optical Gas Analyser (OGA). By employing small, transient variations in gas tensions well within those observed during the normal care of such patients, this approach can provide much more detailed physiological information relating to the lung. By way of example, an increase in end-expiratory lung volume following an inflation manoeuvre can be partitioned between the change relating to the dead space volume and the change relating to the alveolar volume. Furthermore, the measurements also quantify how evenly the lung inflates and deflates during a breathing cycle, and thus changes in ventilation heterogeneity before and after an inflation manoeuvre may also be assessed.

A better understanding of the cardiorespiratory changes that occur in mechanically ventilated patients after a recruitment manoeuvre is performed will aid future studies seeking to determine which patients can benefit from them, when, and why. This will ultimately lead to better medical care and improved ICU survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, aged 18 years or above
* Receiving mechanical ventilation for respiratory failure via an endotracheal tube on ICU

Exclusion Criteria:

* Consultee indicates patient would be likely to decline enrolment
* Patient is receiving palliative care
* Language barriers prevent sufficiently good communication with patient or consultee for full consent to be obtained

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from Intensive Care Units at the Royal Berkshire Hospital in Reading, England. The study population is constituted of patients receiving mechanical ventilation on ICU due to respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional residual capacity | Changes from FRC baseline value measured immediately after PV curve determination and lung recruitment manoeuvre
  To determine whether parameters derived from the airway pressure-volume curve predict changes in static measures of lung volume in response to recruitment manoeuvres

SECONDARY OUTCOMES:
Anatomic dead space | Changes from anatomic dead space baseline value measured immediately after PV curve determination and lung recruitment manoeuvre
  To determine if and how anatomic dead space changes in response to recruitment. manoeuvres
Ventilation inhomogeneity | Changes from ventilation inhomogeneity baseline value measured immediately after PV curve determination and lung recruitment manoeuvre
  To determine if and how ventilatory inhomogeneity changes in response to recruitment manoeuvres. Standard deviation of compliance, dead space, and pulmonary vascular conductance will be used as surrogates of ventilation inhomogeneity.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Robbins, MBBS MA PhD, Study Director — University of Oxford
Locations (1):
- Royal Berkshire Hospital, Royal Berkshire Foundation Trust, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214
- [Background] Esteban A, Frutos-Vivar F, Muriel A, Ferguson ND, Penuelas O, Abraira V, Raymondos K, Rios F, Nin N, Apezteguia C, Violi DA, Thille AW, Brochard L, Gonzalez M, Villagomez AJ, Hurtado J, Davies AR, Du B, Maggiore SM, Pelosi P, Soto L, Tomicic V, D'Empaire G, Matamis D, Abroug F, Moreno RP, Soares MA, Arabi Y, Sandi F, Jibaja M, Amin P, Koh Y, Kuiper MA, Bulow HH, Zeggwagh AA, Anzueto A. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med. 2013 Jul 15;188(2):220-30. doi: 10.1164/rccm.201212-2169OC. PMID 23631814
- [Background] Chiumello D, Carlesso E, Cadringher P, Caironi P, Valenza F, Polli F, Tallarini F, Cozzi P, Cressoni M, Colombo A, Marini JJ, Gattinoni L. Lung stress and strain during mechanical ventilation for acute respiratory distress syndrome. Am J Respir Crit Care Med. 2008 Aug 15;178(4):346-55. doi: 10.1164/rccm.200710-1589OC. Epub 2008 May 1. PMID 18451319
- [Background] Huh JW, Jung H, Choi HS, Hong SB, Lim CM, Koh Y. Efficacy of positive end-expiratory pressure titration after the alveolar recruitment manoeuvre in patients with acute respiratory distress syndrome. Crit Care. 2009;13(1):R22. doi: 10.1186/cc7725. Epub 2009 Feb 24. PMID 19239703
- [Background] Caironi P, Cressoni M, Chiumello D, Ranieri M, Quintel M, Russo SG, Cornejo R, Bugedo G, Carlesso E, Russo R, Caspani L, Gattinoni L. Lung opening and closing during ventilation of acute respiratory distress syndrome. Am J Respir Crit Care Med. 2010 Mar 15;181(6):578-86. doi: 10.1164/rccm.200905-0787OC. Epub 2009 Nov 12. PMID 19910610
- [Background] de Matos GF, Stanzani F, Passos RH, Fontana MF, Albaladejo R, Caserta RE, Santos DC, Borges JB, Amato MB, Barbas CS. How large is the lung recruitability in early acute respiratory distress syndrome: a prospective case series of patients monitored by computed tomography. Crit Care. 2012 Jan 8;16(1):R4. doi: 10.1186/cc10602. PMID 22226331
- [Background] Gattinoni L, Caironi P, Cressoni M, Chiumello D, Ranieri VM, Quintel M, Russo S, Patroniti N, Cornejo R, Bugedo G. Lung recruitment in patients with the acute respiratory distress syndrome. N Engl J Med. 2006 Apr 27;354(17):1775-86. doi: 10.1056/NEJMoa052052. PMID 16641394
- [Background] Gattinoni L, Pelosi P, Suter PM, Pedoto A, Vercesi P, Lissoni A. Acute respiratory distress syndrome caused by pulmonary and extrapulmonary disease. Different syndromes? Am J Respir Crit Care Med. 1998 Jul;158(1):3-11. doi: 10.1164/ajrccm.158.1.9708031. PMID 9655699
- [Background] Vincent JL, Sakr Y, Groeneveld J, Zandstra DF, Hoste E, Malledant Y, Lei K, Sprung CL. ARDS of early or late onset: does it make a difference? Chest. 2010 Jan;137(1):81-7. doi: 10.1378/chest.09-0714. Epub 2009 Oct 9. PMID 19820081
- [Background] Chiumello D, Marino A, Brioni M, Cigada I, Menga F, Colombo A, Crimella F, Algieri I, Cressoni M, Carlesso E, Gattinoni L. Lung Recruitment Assessed by Respiratory Mechanics and Computed Tomography in Patients with Acute Respiratory Distress Syndrome. What Is the Relationship? Am J Respir Crit Care Med. 2016 Jun 1;193(11):1254-63. doi: 10.1164/rccm.201507-1413OC. PMID 26699672
- [Background] Victorino JA, Borges JB, Okamoto VN, Matos GF, Tucci MR, Caramez MP, Tanaka H, Sipmann FS, Santos DC, Barbas CS, Carvalho CR, Amato MB. Imbalances in regional lung ventilation: a validation study on electrical impedance tomography. Am J Respir Crit Care Med. 2004 Apr 1;169(7):791-800. doi: 10.1164/rccm.200301-133OC. Epub 2003 Dec 23. PMID 14693669
- [Background] Luepschen H, Meier T, Grossherr M, Leibecke T, Karsten J, Leonhardt S. Protective ventilation using electrical impedance tomography. Physiol Meas. 2007 Jul;28(7):S247-60. doi: 10.1088/0967-3334/28/7/S18. Epub 2007 Jun 26. PMID 17664639
- [Background] Wrigge H, Zinserling J, Muders T, Varelmann D, Gunther U, von der Groeben C, Magnusson A, Hedenstierna G, Putensen C. Electrical impedance tomography compared with thoracic computed tomography during a slow inflation maneuver in experimental models of lung injury. Crit Care Med. 2008 Mar;36(3):903-9. doi: 10.1097/CCM.0B013E3181652EDD. PMID 18431279
- [Background] Lundin S, Stenqvist O. Electrical impedance tomography: potentials and pitfalls. Curr Opin Crit Care. 2012 Feb;18(1):35-41. doi: 10.1097/MCC.0b013e32834eb462. PMID 22201705
- [Background] Maggiore SM, Jonson B, Richard JC, Jaber S, Lemaire F, Brochard L. Alveolar derecruitment at decremental positive end-expiratory pressure levels in acute lung injury: comparison with the lower inflection point, oxygenation, and compliance. Am J Respir Crit Care Med. 2001 Sep 1;164(5):795-801. doi: 10.1164/ajrccm.164.5.2006071. PMID 11549535
- [Background] Demory D, Arnal JM, Wysocki M, Donati S, Granier I, Corno G, Durand-Gasselin J. Recruitability of the lung estimated by the pressure volume curve hysteresis in ARDS patients. Intensive Care Med. 2008 Nov;34(11):2019-25. doi: 10.1007/s00134-008-1167-8. Epub 2008 Jun 25. PMID 18575846
- [Background] Arnal JM, Paquet J, Wysocki M, Demory D, Donati S, Granier I, Corno G, Durand-Gasselin J. Optimal duration of a sustained inflation recruitment maneuver in ARDS patients. Intensive Care Med. 2011 Oct;37(10):1588-94. doi: 10.1007/s00134-011-2323-0. Epub 2011 Aug 20. PMID 21858522
- [Background] Chen L, Del Sorbo L, Grieco DL, Junhasavasdikul D, Rittayamai N, Soliman I, Sklar MC, Rauseo M, Ferguson ND, Fan E, Richard JM, Brochard L. Potential for Lung Recruitment Estimated by the Recruitment-to-Inflation Ratio in Acute Respiratory Distress Syndrome. A Clinical Trial. Am J Respir Crit Care Med. 2020 Jan 15;201(2):178-187. doi: 10.1164/rccm.201902-0334OC. PMID 31577153
- [Background] Papazian L, Aubron C, Brochard L, Chiche JD, Combes A, Dreyfuss D, Forel JM, Guerin C, Jaber S, Mekontso-Dessap A, Mercat A, Richard JC, Roux D, Vieillard-Baron A, Faure H. Formal guidelines: management of acute respiratory distress syndrome. Ann Intensive Care. 2019 Jun 13;9(1):69. doi: 10.1186/s13613-019-0540-9. PMID 31197492